CLINICAL TRIAL: NCT03155737
Title: Self-administered Acupressure for Knee Osteoarthritis in Middle- and Older Adults: A Pilot Randomized Controlled Trial
Brief Title: Self-administered Acupressure for Knee Osteoarthritis: A Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AcupKneeOA
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-acupressure Training (Experimental): Subjects in the self-administered acupressure exercise group will receive two 1.5 hours acupressure training sessions. The training will be conducted in a group format with 4-7 subjects per group. Each subject will then receive a handout and an acupressure log. The handout includes a picture-illustrating acupressure step-by-step protocol. They will be told to perform the self-acupressure twice per day for 6 weeks.
  Interventions: Other: Self-acupressure
- Knee Health Education (Active Comparator): Subjects in the health education control group will receive knowledge related to knee OA. The health education will be conducted in a talk format for 1.5 hours for two sessions.
  Interventions: Other: Knee health education

INTERVENTIONS:
Other: Self-acupressure — A training course will be offered to subjects in this group to train them to perform self-acupressure.
  Arms: Self-acupressure Training
Other: Knee health education — A course regarding knee health will be offered to the subjects in this group.
  Arms: Knee Health Education

SUMMARY:
Objectives: To test the feasibility of the study design and clinical effects of self-administered acupressure on relieving knee osteoarthritis (OA) pain.

Hypothesis: self-administered acupressure would have a superior beneficial effect compared to health education control group in terms of pain relief in patients with knee osteoarthritis across the 6-week study period.

Design and subjects: A pilot randomized controlled trial. 36 subjects with knee OA will be recruited; 18 per group. All eligible subjects will be randomized to either self-administered acupressure or health education control group in 1:1 ratio.

Interventions: Subjects in the self-acupressure group will attend two 1.5 hours training sessions to learn self-acupressure and will practice self-acupressure every morning and night for 6 weeks; subjects in the education control group will receive two 1.5 hours training sessions to learn the health information related to knee OA.

Main outcome measures: The primary outcome measure is the numerical rating scale for knee pain. Other measures include Western Ontario and McMaster University Osteoarthritis Index, knees' range of motion (ROM), and SF-6D. Acceptability of the self-acupressure training course will also be evaluated.

Data Analysis: Differences in the questionnaire scores and ROM will be examined using a mixed-effects model. Both completer and intention-to-treat analyses will be conducted. Effect sizes will be computed by dividing the difference in means by the pooled standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* ethnic Chinese;
* aged 50 -70 years
* fulfills any 3 of the following criteria proposed by Altman et al., (1986): ( I. morning stiffness</= 30 min; ii. crepitus on active joint motion; iii. bone tenderness; iv. bone enlargement; or v. no palpable joint warmth);
* having knee pain for at least 3 months;
* ability to provide informed consent;
* ability to comprehend Chinese; and
* Knee pain ≥3/10 and </= 7 on a Likert pain scale from 1-10

Exclusion Criteria:

* medical diagnoses or conditions that preclude individuals from active participation (bleeding disorders, alcohol or drug abuse);
* presence of skin lesions or infections at the treatment sites;
* currently participating in other interventional research studies for knee OA;
* cognitive impairment preventing informed consent or understanding of instructions
* body mass index over 25, the obese criteria for Asians (Anuurad et al., 2003);
* knee pain related to other conditions (cancer, fracture, rheumatoid arthritis, rheumatism) as screened according to the red flags for further investigation or referral in the NICE 2014 Guidelines for Osteoarthritis of the knee;
* had previous foot injury or trauma;
* using of steroid for knee pain;
* pregnancy or contemplating pregnancy;
* ever received acupressure for knee OA over the past 6 months.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Pain severity numerical rating scale | Week 6
  A single 11-point numeric scale ranges from 0 to 10 in 1 cm intervals (zero: no pain, 10: greatest pain imaginable).

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Baseline, Week 2, Week 4, Week 6
  The Western and McMaster Universities Osteoarthritis Index (WOMAC, Likert version 3.1) covered pain, physical function, and stiffness related to knee osteoarthritis. The physical function subscale (consisting of 17 items) will be adopted to assess the level of physical function in patients with knee osteoarthritis under different activities.
Range of motion (ROM) | Baseline, Week 6
  Range of motion is recorded in degrees by using a goniometer. ROM can be used to address the inter-relationship between ROMs of joint action and disability in patient with knee OA.
Short Form 6D (SF-6D) | Baseline, Week 6
  The Short Form -6D is a preference-based measure of health derived from a selection of SF-36 items for economic evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No